CLINICAL TRIAL: NCT04311528
Title: Immunogenicity, Compliance, Knowledge and Attitudes in Postpartum Women During a Two Dose 9-valent HPV Vaccination Series
Brief Title: 9-valent HPV Vaccine in Postpartum Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PP-HPV
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Human Papilloma Virus

STUDY DESIGN:
Intervention Model Description: open label; all subjects will receive the 9-valent HPV vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: 9-valent HPV vaccine — 9-valent HPV vaccine

SUMMARY:
This study will evaluate the immunogenicity of the 9-valent HPV vaccine in post-partum women age 16-45.

DETAILED DESCRIPTION:
Women age 16-45 who are pregnant or who have just delivered will be eligible to participate in a study involving the 9-valent HPV vaccine. For clarification, women who are pregnant are eligible to sign consent, but the first vaccine will not occur until after delivery. Vaccine # 1 must occur within seven days of delivery.

The main objective of the study is to determine the immunogenicity of the vaccine in postpartum women. The immunogenicity results will be compared to that of non-postpartum women of the same age, 16-45.

Women will participate for approximately 12 months and will complete a total of 4 visits during that time frame.

ELIGIBILITY:
Inclusion Criteria:

* Female between the ages of 16 and 45 years of age at enrollment
* Postpartum (Day 1 vaccination to occur within 1 week of delivery)
* Judged to be in good health on the basis of medical history and physical examination
* Able to fully understand study procedures, alternative treatments available, the risks involved in the study and voluntarily agrees to participate by giving written informed consent
* Able to read, understand, and complete the questionnaires

Exclusion Criteria:

* Has a known allergy to any vaccine component, including aluminum, yeast, or BENZONASE™
* Has thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections
* Is currently immunocompromised or has been diagnosed as having a congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition.
* Is receiving or has received in the year prior to enrollment the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide, TNF-α antagonists, monoclonal antibody therapies (including rituximab), intravenous gamma globulin (IVIG), antilymphocyte sera, or other therapy known to interfere with the immune response. With regard to systemic corticosteroids, a subject will be excluded if she is currently receiving steroid therapy, has recently (within 2 weeks of enrollment) received such therapy, or has received 2 or more courses of high dose corticosteroids (orally or parenterally) lasting at least 1 week in duration in the year prior to enrollment. The use of inhaled, nasal, or topical steroids are considered eligible for the study
* Has received any immune globulin product (including RhoGAM™) or other blood- derived product within 3 months prior to Day 1 vaccination or plans to receive such product during the study
* Has received a marketed HPV vaccine
* Has had a fever of > 100° within 24-hour period prior to the Day 1 vaccination

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — study is specifically to test the immunogenicity of postpartum women, therefore, only females will be eligible to participate
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer | Day 0, Month 7 and Month 12
  immunogenicity testing using 9-plex competitive Luminex Immuno Assay (9-plex cLIA)